CLINICAL TRIAL: NCT02595697
Title: An Efficacy Trail of Enhanced Milieu Teaching Language Intervention Plus Joint Attention, Engagement, Regulation Intervention for Toddlers With Autism
Brief Title: Communication Intervention for Toddlers With Autism
Acronym: J-EMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, Ann Kaiser, Ann P Kaiser, PhD, Vanderbilt University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: R324A150094
Record Dates: First submitted 2015-10-02; First posted 2015-11-03 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- J-EMT for Toddlers with Autism (Experimental): The J-EMT intervention:(a) teach foundational social communicative behaviors, (b) teach related skills that predict long term language outcomes, (c) teach a range of communicative functions, (d) target specific spoken language skills as well as foundational skills, (e) incorporate instructional methods, contexts, and partners that increase social use of language in natural contexts, and (f) promote generalization and maintenance of newly learned skills to everyday activities and routines. In addition, because parents are essential partners for young children with ASD who are learning to communicate, studies are needed that (g) include parents and (h) specify the method and fidelity of parent instruction and fidelity and dosage with which parents use the trained strategies
  Interventions: Behavioral: J-EMT for Toddlers with Autism
- Business as Usual Control Group (No Intervention): All children, regardless of group assignment will participate in all assessments. Children randomized to the control group will not receive intervention, but will complete all other research procedures. Other treatments that all children receive in the community will be recorded with bi-monthly surveys.

INTERVENTIONS:
Behavioral: J-EMT for Toddlers with Autism — Children assigned to the J-EMT group will receive a total of 48, 1-hour direct intervention sessions over six months that will include teaching their parents to implement J-EMT procedures across daily activities.
  Other Names: Communication Intervention for Toddlers with Autism
  Arms: J-EMT for Toddlers with Autism

SUMMARY:
The goal of this study is to conduct an efficacy trial to determine whether an early communication intervention which blends two evidence-based interventions, Enhanced Milieu Teaching (EMT) and Joint Attention, Symbolic Play and Regulation Intervention (JASPER), improves social communication in toddlers with Autism Spectrum Disorder (ASD).

DETAILED DESCRIPTION:
This study tests the blended intervention (J-EMT) in a parent-plus-therapist-implementation model that has been demonstrated to be effective with other populations.

The J-EMT communication intervention is tailored to the specific social communication characteristics of children with ASD and is delivered during a critical period in early communication development for these children.

In this study, the investigators compare this blended intervention (J-EMT) to a business as usual (BAU) comparison group. Children assigned to the J-EMT group will receive a total of 48, 1-hour direct intervention sessions over six months that will include teaching their parents to implement J-EMT procedures across daily activities.

The investigators will examine social communication and child vocalizations, expressive and receptive language, symbolic play, and symbol-infused joint engagement to determine whether J-EMT changes both a primary functional outcome and the underlying specific skills that contribute to effective social communication in children with ASD.

Results from this study will indicate the efficacy of this variation of parent-plus-therapist-implemented EMT (i.e., J-EMT) specifically tailored to the characteristics of young children with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Between 24 and 36 months of age
* A diagnosis of ASD as confirmed by the ADOS-2 (module 1)
* Signed informed consent
* Parent willing to be trained

Exclusion Criteria:

* Other diagnosis or disability
* Abnormal hearing and/or vision
* Language other than English is the primary language spoken at home

Ages: 24 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2015-07; Primary Completion 2019-12 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Number of spontaneous social communication attempts made as assessed by a 20 minute lanugage sample. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ann P Kaiser, PhD, Principal Investigator — Vanderbilt University
Locations (2):
- United States (2):
  - Northwestern University, Evanston, Illinois
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Roberts MY, Stern YS, Grauzer J, Nietfeld J, Thompson S, Jones M, Kaat AJ, Kaiser AP. Teaching Caregivers to Support Social Communication: Results From a Randomized Clinical Trial of Autistic Toddlers. Am J Speech Lang Pathol. 2023 Jan 11;32(1):115-127. doi: 10.1044/2022_AJSLP-22-00133. Epub 2022 Dec 16. PMID 36525627